CLINICAL TRIAL: NCT07038096
Title: A Phase Ib/II Study of the Tolerability, Safety, Efficacy, and Pharmacokinetics of ZG006 in Combination With ZG005 in Participants With Advanced Small Cell Lung Cancer or Neuroendocrine Carcinoma(NEC)
Brief Title: ZG006 and ZG005 in Participants With Small Cell Lung Cancer or Neuroendocrine Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZG006-ZG005-001
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer; Neuroendocrine Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma; Carcinoma, Neuroendocrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ib: Part1-Dose Escalation (Experimental): This study will employ the traditional "3+3" dose escalation design. Ultimately, two combination dosing cohorts will be selected to enter Part 2, the dose expansion phase, based on a comprehensive evaluation of the safety and pharmacokinetic (PK) data obtained by the investigators and the sponsor.
  Interventions: Drug: ZG006; Drug: ZG005
- Phase Ib: Part2-Dose Expansion (Experimental): The safety and pharmacokinetic (PK) data obtained in Part 1 will be used to determine two expansion phase doses of the ZG006 and ZG005 combination. The dose expansion study will further evaluate the efficacy of the two selected combination dosing cohorts in patients with advanced small cell lung cancer and neuroendocrine carcinoma.
  Interventions: Drug: ZG006; Drug: ZG005
- Phase II (Experimental): Participants will receive the RP2D of ZG006 in combination with ZG005 identified in Phase Ib of the study.
  Interventions: Drug: ZG006; Drug: ZG005

INTERVENTIONS:
Drug: ZG006 — ZG006 will be administered as an intravenous (IV) infusion.
Drug: ZG005 — ZG005 will be administered as an intravenous (IV) infusion.

SUMMARY:
This study is a randomized, multicenter, Phase Ib/II clinical trial, aimed at evaluating the efficacy and safety of the combination of ZG006 and ZG005 in patients with advanced small cell lung cancer and neuroendocrine carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Fully understand the study and voluntarily sign the informed consent form.
* Male or female 18-70 years of age.
* Participants with advanced small cell lung cancer or neuroendocrine carcinoma confirmed by histopathology or cytology.
* Eastern Cooperative Oncology Group (ECOG) 0 to 1.
* Life expectancy > 3 months.

Exclusion Criteria:

* The investigator believes that the subject has other reasons that make them unsuitable for participation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Dose-limiting Toxicity (DLT) | up to 28 days
Number of Participants With Treatment-emergent Adverse Events (TEAEs) | Up to 2 years
Objective Response Rate (ORR) | Up to 2 years
  The objective response rate was defined as the percentage of participants with a confirmed best overall response of complete response (CR) or partial response (PR) based on the modified RECIST v1.1.

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 2 years
Disease Control Rate (DCR) | Up to 2 years
Progression-free Survival (PFS) | Up to 2 years
Overall Survival (OS) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China